CLINICAL TRIAL: NCT05874310
Title: An Open-label, Single-center, Dose-escalation Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Intraocular Administration of FT-002 in Subjects With RPGR Mutation-associated X-linked Retinitis Pigmentosa.
Brief Title: Gene Therapy for Subjects With RPGR Mutation-associated X-linked Retinitis Pigmentosa
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other); Peking Union Medical College Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT002RP-1
Record Dates: First submitted 2023-04-29; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-08

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: X-linked retinitis pigmentosa patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose FT-002 (Experimental): Intraocular injection of a single low dose of FT-002
  Interventions: Genetic: FT-002
- Intermediate dose FT-002 (Experimental): Intraocular injection of a single Intermediate dose of FT-002
  Interventions: Genetic: FT-002
- High dose FT-002 (Experimental): Intraocular injection of a single High dose of FT-002
  Interventions: Genetic: FT-002

INTERVENTIONS:
Genetic: FT-002 — Comparison of different dosages of FT-002

SUMMARY:
A clinical trial of gene therapy for patients with X-linked retinitis pigmentosa (XLRP).

ELIGIBILITY:
Inclusion Criteria:

1.Subjects that are willing and able to follow study procedures; 2.Males aged 8-45 years old at the time of signing the Informed Consent Form; 4.Subjects who are confirmed with variants of RPGR ;

Exclusion Criteria:

1.Have other retinal degenerative diseases, such as retinal degeneration caused by other known Inherited retinal disease gene variants or previously received an gene therapy product.

Ages: 8 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | from FT-002 administration through up to 1 years
  Number and proportion of Adverse Events

SECONDARY OUTCOMES:
Change in visual function | from FT-002 administration through up to 1 years
  Change in retinal function as assessed by mean retinal sensitivity within the 30-degree visual field
Change in retinal structure as assessed by Optical Coherence Tomography | from FT-002 administration through up to 1 years
  Change in Outer Nuclear Layer Thickness from baseline as assessed by Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Gezhi Xu, Principal Investigator — Eye & ENT Hospital of Fudan University; Ruifang Sui, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Eye & ENT hospital of Fudan university, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Researchers qualified can request the dataset, including de-identified individual subject data.